CLINICAL TRIAL: NCT07174986
Title: "A Randomized Trial Assessing the Effect of Early Double Sequential Defibrillation With Anterior-posterior and Anterior Lateral Pad Placement and Sequential Defibrillation Compared to Standard Pad Placement and Single Defibrillation in Patients With Out of Hospital Cardiac Arrest With Initial Shockable Rhythm and at Least One Failed Standard Defibrillation"
Brief Title: Early Double Sequential Defibrillation in Out of Hospital Cardiac Arrest
Acronym: DOUBLE D
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gabriel Riva (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Region Stockholm (Other Government); Vastra Gotaland Region (Other Government); Region Halland (Other); Laerdal Foundation (Other)
Responsible Party: Sponsor-Investigator, Gabriel Riva, Principal Investigator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIV-ID-25-01-051015; Dnr 2025-03532-01 (Other: Swedish etical review authority)
Record Dates: First submitted 2025-09-03; First posted 2025-09-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Out of Hospital Cardiac Arrest; Ventricular Fibrillation; Defibrillation; CPR; ACLS; Sudden Death
Keywords: Double sequential defibrillation; Double sequential external defibrillation; ACLS
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation; Death, Sudden

STUDY DESIGN:
Intervention Model Description: Academic, investigator initiated, open-label pilot study with a randomized controlled trial (RCT) design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Double sequential defibrillation (Experimental): If the patient is randomized to the DSD group, the ambulance crew team will apply the second defibrillator with electrodes placed in the A-P position as soon as possible.
  Defibrillation is performed by one person defibrillating both defibrillators in a sequential manner "Double Sequential Defibrillation" (DSD). All consecutive defibrillations will thereafter be performed with the DSD strategy until ROSC, termination of resuscitation or decision to move the patient to hospital.
  Interventions: Device: Double sequential defibirllation
- Standard defibrillation (Active Comparator): If the patient is randomized to the standard defibrillation group, the ambulance crew team will continue Advanced life support in accordance with standard of care and continue to perform standard defibibrillation using one defibrillator. All consecutive defibrillations will thereafter be performed with the standard defibrillation strategy until ROSC, termination of resuscitation or decision to move the patient to hospital.
  Interventions: Device: Standard defibrillation

INTERVENTIONS:
Device: Double sequential defibirllation — A second defibrillator will be applyed with electrodes placed in the A-P position and defibrillation will be performed with two defibrllators in a sequential manner
  Other Names: DSD
  Arms: Early Double sequential defibrillation
Device: Standard defibrillation — Standard defibrillation uning one defibrillator
  Arms: Standard defibrillation

SUMMARY:
Some of the patients affected by Out-of-hospital cardiac arrest (OHCA) with ventricular fibrillation (VF)/ventricular tachycardia (VT) do not respond to initial defibrillation. The survival decreases with number of defibrillations required to terminate VF/VT. In 2022, one prospective cluster randomized trial showed increased survival among (OHCA) patients in refractory VF using Double Sequential Defibrillation (DSD). If DSD can increase survival among all patients in VF that dont respond to one defibrillation, i.e. before it has become refractory is not known.

The aim of this trial is to assess survival with a double defibrillation strategy initiated as soon as possible among patients with Out of Hospital Cardiac Arrest with initial shockable rhythm and at least one failed standard defibrillation, compared with continued resuscitation using standard defibrillation.

DETAILED DESCRIPTION:
Background: Out-of-hospital cardiac arrest (OHCA) affects about 270,000 individuals in Europe annually.[1] In OHCA, presenting with ventricular fibrillation (VF) or pulseless ventricular tachycardia (VT) amendable to defibrillation are among the strongest predictors of survival.[2] If defibrillation can be done successfully within the first 3-5 minutes survival can be as high as 70 %.[3] However, some patients in VT/VF do not respond to initial defibrillation, and survival decreases with number of defibrillations required to terminate VT/VF.[4]

In 2022, one prospective cluster randomized trial showed increased survival among OHCA patients in refractory VF using an alternative defibrillation strategy with either, switching to Anterior-Posterior defibrillation pad placements (A-P) or Double Sequential Defibrillation "DSD", (Using two defibrillators, one in the standard anterior-lateral position (A-L) and one in A-P position and defibrillation in rapid sequence) compared to standard defibrillation pad placement.[5] Refractory VF was defined as VF that persisted despite three consecutive defibrillations with defibrillation pads in the standard position.

These results prompted the International Liaison Committee on Resuscitation (ILCOR) to release a statement of treatment recommendation on DSD in March 6, 2023. It suggested that "…either vector change or DSD may be considered for adults with cardiac arrest who remain in VF or pulseless VT despite three defibrillations (weak recommendation, low certainty of evidence)." [6] Further, if DSD would be used it should be performed with a methodology similar to that described in the trial by Cheskes et al.

However, several questions remain. Knowledge gaps highlighted in the ILCOR statement included if the results from this one cluster randomized trial could be reproduced in any other setting. Further, since survival is inversely associated with the number of defibrillation shocks, if earlier application of DSD could lead to even higher survival for patients not in refractory VF has never been studied.

Study rationale: In order to evaluate if an early DSD-strategy could benefit all patients with VT/VF after the first shock, including those not in refractory VF, the Double-D trial is designed. If DSD would prove to be superior to standard defibrillation in a broader cardiac arrest population, also among those not in refractory VF, this would have a large impact on how Advanced Cardiac Life Support (ACLS) should be performed.

Design: This is an academic, investigator initiated, open-label pilot study with a randomized controlled trial (RCT) design and 1:1 allocation (1 DSD: 1 standard). Screening for inclusion will be performed in all cardiac arrests by participating EMS units where there are two study-specific defibrillators available on site.

Study population: Adult OHCA patients with pulseless VT/VF at initial rhythm analysis, at least one defibrillation performed in standard A-L position without return of spontaneous circulation (ROSC).

P: Adult patients, 18 years or older, with OHCA, initial shockable rhythm (VT/VF) and, at least, one defibrillation performed in standard position and ongoing CPR (no ROSC).

I: Application of a second defibrillator with pad-placement in the anterior-posterior (A-P) position as early as possible after the first shock and double sequential defibrillation after the following rhythm analysis if the patient is still in VT/VF.

C: Standard defibrillation electrode placement (A-L) and routine defibrillation with one defibrillator after the following rhythm analysis if the patient is still in VT/VF.

O: Primary outcome is 30-day survival.

The trial will be conducted by participating ambulance units attending OHCA´s. These units will perform screening for inclusion, randomization, intervention or control treatment and initial follow up.

ELIGIBILITY:
Inclusion Criteria:

* OHCA patients with VT/VF at first rhythm analysis and at least one defibrillation performed in standard (A-L) position

Exclusion Criteria:

* Age < 18 years
* Obvious pregnancy
* Known preexisting Do Not Attempt Resuscitation order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 916 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
30 day survival | 30 days
  Survival at 30 days

SECONDARY OUTCOMES:
Neurological function at hospital discharge, mRS (modified Ranking scale, 1-6 where 1 indicates better function) | 30 days
  Neurological function at hospital discharge (mRS)
Survival to hospital Admission | 1 day
  Admitted alive to a hospital ward
Survival to hospital discharge | 30 days
  Discharged alive from hospital
90 days survival | 90 days
  Survival to 90 days

OTHER OUTCOMES:
Neurological function at 90 days (mRS) | 90 days
  Neurological function at 90 days (modified Ranking scale)
Neurological function at 180 days (mRS) | 180 days
  Neurological function (modified Ranking Scale)
ROSC | 1 day
  Proportion of patients with sustained return of spontaneous circulation (ROSC) at hospital arrival
Number of defibrillations to sustained ROSC | 1 day
  Total number of defibrillations to sustained ROSC
Termination of ventricular fibrillation | 1 day
  Termination of ventricular fibrillation
Helath related quality of life at 90 days | 90 days
  Helath related quality of life at 90 days
Health related quality of life at 180 days | 180 days
  Health related quality of life at 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Riva, M.D. Ph.D., Study Director — Center for resuscitation Science. Department of clinical sience and education. Södersjukhuset, Karolinksa Institutet, Stockholm, Sweden; Akil Awad, M.D. Ph.D., Principal Investigator — Center for resuscitation Science. Department of clinical sience and education. Södersjukhuset, Karolinksa Institutet, Stockholm, Sweden; Carl Magnusson, R.N., Ph.D., Study Chair — Shalgrenska University Hospital; Andreas Claesson, R.N. Ph.D., Study Chair — Center for resuscitation Science. Department of clinical sience and education. Södersjukhuset, Karolinksa Institutet, Stockholm, Sweden; Johan Israelsson, R.N. Ph.D., Study Chair — ICARE, Department of Health and Caring Sciences, Linnaeus University
Locations (8):
- Sweden (8):
  - Ambulanssjukvården, Region Halland, Halmstad, Halland County
  - Ambulanssjukvården Region Värmland, Karlstad, Värmland County
  - Sjukvården i väster, Alingsås
  - Emergency medical services, Södra Älvsborgs Sjukhus, Region Västra Götaland, Borås
  - Prehospital Intensive Care Unit (PIV) AnOPIVA Östra Sjukhuset/SU, Gothenburg
  - Shalgrenska University Hospital, Gothenburg
  - Ambulanssjukvården Skaraborgs Sjukhus, Västra Götalandsregionen (SKAS), Skövde
  - Emergency medical services NU-Sjukvården, Region Västra Götaland, Trollhättan